#### **Statistical Analysis Plan Version 5**

**Study ID:** 213403

**Study Official Title:** A Randomized, Phase 2, Double-blind Study to Evaluate the Efficacy of Dostarlimab Plus Chemotherapy Versus Pembrolizumab Plus Chemotherapy in Metastatic Non-Squamous Non-Small Cell Lung Cancer

**NCT ID:** NCT04581824

**Date of Document:** 22-Aug-2024

**Division** : Worldwide Development

**Information Type** : Statistical Analysis Plan (SAP)

#### **Title Page**

**Protocol Title:** A Randomized, Phase 2, Double-blind Study to Evaluate the

Efficacy of Dostarlimab Plus Chemotherapy versus

Pembrolizumab Plus Chemotherapy in Metastatic Non-Squamous

Non-Small Cell Lung Cancer

**Protocol Number:** 213403

Compound Number: GSK4057190 (Dostarlimab)

**Short Title:** Efficacy Comparison of Dostarlimab Plus Chemotherapy vs

Pembrolizumab Plus Chemotherapy in Participants with Metastatic

Non-squamous Non-small Cell Lung Cancer

Acronym: PERLA

**Sponsor Name:** GlaxoSmithKline Research & Development Limited

#### **Regulatory Agency Identifier Number(s)**

**Registry** ID

*IND Number* 150997

*EudraCT* 2020-002327-11

Number

#### **SAP Author(s):**

# PPD Principal Statistician, Study Lead Statistician, Development Biostatistics Oncology PPD Statistician, Veramed PPD Senior Statistician, Veramed

#### **SAP Team Review Confirmations (Veeva Vault Confirmation):**



#### SAP Biostatistics Line Approval (Pharma TMF eSignature):



Copyright 2024 the GlaxoSmithKline group of companies. All rights reserved. Unauthorized copying or use of this information is prohibited.

# TABLE OF CONTENTS

| | | | | l | PAGE |
|---|---|---|---|---|---|
| VE | RSION | HISTORY | | | 6 |
| 1. | INTRO | | J | | 13 |
| 1. | 1.1. | Objective | s, Estimands | and Endpoints | 13 |
| | | 1.1.1.<br>1.1.2. | | d Endpoints | |
| | 1.2. | | | | |
| 2. | STAT | ISTICAL H | VPOTHESES. | | 18 |
| ۷. | 2.1. | | | | |
| 3. | ANAL | YSIS SETS | 3 | | 19 |
| 4. | | | | | |
| | 4.1. | | | S | |
| | | 4.1.1. | | odology | |
| | | 4.1.2. | | nition | |
| | | 4.1.3. | | tudies | |
| | | 4.1.4. | | <b>3</b> | |
| | | 4.1.5. | | tion Summaries | |
| | 4.2. | Primary E | | /ses | |
| | | 4.2.1. | | endpoint | |
| | | 4.2.2. | Main analytic | al approach | 22 |
| | | 4.2.3. | Sensitivity an | alyses | 23 |
| | 4.3. | Seconda | ry Endpoints A | Analyses | 23 |
| | | 4.3.1. | | endpoints | |
| | | | 4.3.1.1. Ov | verall Survival (OS) | 23 |
| | | | 4.3.1.2. Pr | ogression-Free Survival per RECIST v1.1<br>FS) | |
| | | 4.3.2. | | al approach | |
| | | 4.0.2. | | verall Survival (OS) | |
| | | | 4.3.2.2. Pr | ogression-Free Survival per RECIST v1.1 | |
| | | | | FS) | |
| | 4.4. | | e Secondary | Endpoint(s) | |
| | | 4.4.1. | | nts/Serious Adverse Events | |
| | | | 4.4.1.1. Ac | Iverse Events of Special Interest | 28 |

Statistical Analysis Plan 213403 V5 4.7. Interim Analyses .......40 4.8. SAMPLE SIZE DETERMINATION ......41 SUPPORTING DOCUMENTATION ......41 Appendix 1 Abbreviations and Trademarks......41 6.1.1. List of Abbreviations ......41 Trademarks .......43 6.1.2.

#### Statistical Analysis Plan 213403 V5

# **LIST OF TABLES**

| PAGE |
|--------------------------------------------|
| Table 1 SAP Version History Summary |
| Table 2 Estimands |
| Table 3 Analysis Sets |
| CI |
| Table 6 Adverse Events of Special Interest |

# **VERSION HISTORY**

Table 1 SAP Version History Summary

| SAP<br>Version | Document<br>Date | Protocol Version (Date) on which SAP is Based | Change | Rationale |
|---|---|---|---|---|
| 1 | 15 March<br>2022 | Version 04 30 November 2021 | Not Applicable | Original version |
| 2 | 27 July<br>2022 | Version 04 30 November 2021 | ICCI | CCI |

| SAP<br>Version | Document<br>Date | Protocol Version (Date) on which SAP is Based | Change | Rationale |
|---|---|---|---|---|
| 3 | 07 June 2023 | Version 05 14 February 2023 | CCI | CCI |

| 4 16 April 2024 Version 05 14 February 2023 | SAP<br>Version | Document<br>Date | Protocol Version (Date) on which SAP is Based | Change | Rationale |
|---|---|---|---|---|---|
| | 4 | 16 April 2024 | Version 05<br>14 February | CCI | |

| SAP<br>Version | Document<br>Date | Protocol<br>Version<br>(Date) on<br>which SAP<br>is Based | Change | Rationale |
|---|---|---|---|---|
| | | | CCI | CCI |

| SAP<br>Version | Document<br>Date | Protocol<br>Version<br>(Date) on<br>which SAP<br>is Based | Change | Rationale |
|---|---|---|---|---|
| | | | CCI | CCI |

| SAP<br>Version | Document<br>Date | Protocol<br>Version<br>(Date) on<br>which SAP<br>is Based | Change | Rationale |
|---|---|---|---|---|
| | | | CCI | CCI |
| 5 | 22 Av. | Various 05 | _ | |
| 5 | 22 Aug<br>2024 | Version 05<br>14 February<br>2024 | | |

| SAP<br>Version | Document<br>Date | Protocol<br>Version<br>(Date) on<br>which SAP<br>is Based | Change | Rationale |
|---|---|---|---|---|
| | | | CCI | CCI |

#### 1. INTRODUCTION

The purpose of this SAP is to describe the planned analyses to be included in the Clinical Study Report for Study 213403 (PERLA). Details of the final analyses are provided.

Descriptive study population analyses such as summary of demography and baseline characteristics and additional detail with regards to data handling conventions and the specification of data displays will be provided in the Output and Programming Specification (OPS) document.

# 1.1. Objectives, Estimands and Endpoints

# 1.1.1. Objectives and Endpoints

| | Endpoints |
|---|---|
| Primary | |
| To compare the ORR of PD1 inhibitor dostarlimab vs pembrolizumab administered in combination with chemotherapy as evaluated using RECIST v1.1 based on BICR in participants with metastatic nonsquamous NSCLC, without a known EGFR, ALK, ROS1, or BRAF V600E mutation or other genomic aberration for which an approved targeted therapy is available, who have received no prior treatment of metastatic disease | The primary efficacy endpoint ORR will be evaluated by RECIST v1.1 based on BICR and will be defined as the proportion of participants with BOR of CR or PR in the analysis population. |
| Secondary | |
| To evaluate the following measures of clinical<br>benefit of PD-1 inhibitor administered in | OS will be defined as the time from the date of<br>randomization to the date of death by any cause. |
| combination with chemotherapy: OS PFS evaluated using RECIST v1.1 based on Investigator assessment | <ul> <li>PFS will be evaluated using RECIST v1.1 based<br/>on Investigator assessment and will be defined as<br/>the time from the date of randomization to the<br/>date of PD or death by any cause, whichever<br/>occurs first.</li> </ul> |
| To evaluate the safety of PD-1 inhibitor in combination with chemotherapy | Assess the incidence of TEAEs, SAEs, irAEs, TEAEs leading to death, and AEs leading to discontinuation occurring while participants are on treatment or up to 90 days after the last dose of study treatment. Clinical laboratory parameters (hematology, chemistry, thyroid function, urinalysis), vital signs, ECOG performance status, ECG parameters, physical examinations, and usage of concomitant medications will be collected. |
| Exploratory | |





#### Table 2 Estimands

| | | Estimand | | | |
|---|---|---|---|---|---|
| Objective | Estimand<br>Category | Population | Variable/<br>Endpoint | Intercurrent Event<br>Strategy | Population<br>Level<br>Summary<br>Measure |
| Primary Objective: | | | | | |
| To compare the ORR of dostarlimab vs pembrolizumab administered in combination with chemotherapy as evaluated using RECIST v1.1 based on BICR in participants with metastatic nonsquamous NSCLC, without a known EGFR, ALK, ROS-1, or BRAF V600E mutation or other genomic aberration for which an approved targeted | Primary | Participants with metastatic non-squamous NSCLC, without a known EGFR, ALK, ROS-1, or BRAF V600E mutation or other genomic aberration for which an approved targeted therapy is available, who have received no prior treatment of metastatic disease | ORR | CCI | |

| | | Estimand | | | |
|---|---|---|---|---|---|
| Objective | Estimand<br>Category | Population | Variable/<br>Endpoint | Intercurrent Event<br>Strategy | Population<br>Level<br>Summary<br>Measure |
| therapy is available,<br>who have received<br>no prior treatment of<br>metastatic disease | | | | | |

#### 1.2. Study Design



Abbreviations: 1L=first-line; NSCLC=non-small cell lung cancer.

Note: Both arms will be stratified by PD-L1 status (TPS <1% vs 1% to 49% vs ≥50%) and smoking status (never vs former/current)

#### **Design Features**

- This is a randomized, Phase 2, double-blind, 2-arm study to compare the efficacy and safety of PD-1 inhibitors dostarlimab and pembrolizumab, when administered in combination with chemotherapy, in male and female participants 18 years and older with non-squamous NSCLC without a known sensitizing epidermal growth factor receptor (EGFR), anaplastic lymphoma kinase (ALK), receptor tyrosine kinase-1 (ROS-1), or proto-oncogene B-raf (BRAF) V600E mutation or other genomic aberration for which an approved targeted therapy is available who have not received previous systemic anticancer therapy for metastatic disease.
- Approximately 240 participants will be randomized in a 1:1 ratio into the
  dostarlimab plus chemotherapy arm or the pembrolizumab plus
  chemotherapy arm, such that approximately 120 evaluable participants
  in each of the 2 arms complete the study.
- Randomization will be stratified by:
  - PD-L1 status of the tumor (TPS <1% versus 1% to 49% versus ≥50%);</li>

#### **Overview of Study Design and Key Features** Smoking status (never versus former/current). 0 The study consists of a Screening Period (Day -28 to Day -1) for completion of all Screening assessments and subsequent randomization, a Treatment Period, an EOT Visit (within 7 days of the decision to discontinue treatment for any reason), a Safety Follow-up Period with a visit at 30 (+7) and 90 (+7) days after the last dose of study treatment, and a Post-treatment Follow-up Period with assessments occurring 180 days after the last dose of study treatment and every 90 (±14) days thereafter, continuing until death, withdrawal of consent, or the end of study data collection. The study will last approximately 5 years. During the Treatment Period participants will take part in up to 35 cycles with a visit frequency of Q3W (cycles are 21 [±3] days). Study Dostarlimab will be administered through a 30-minute infusion at a intervention dose of 500 mg IV Q3W up to a maximum of 35 cycles total (approximately 24 months). Pembrolizumab will be administered through a 30-minute infusion at a dose of 200 mg Q3W up to a maximum of 35 cycles total (approximately 24 months). Chemotherapy (standard of care) will be administered to participants in both treatment arms: Pemetrexed will be administered at 500 mg/m2 IV through a 10minute IV infusion Q3W, up to a maximum of 35 cycles total (approximately 24 months). Platinum chemotherapy (Cisplatin / Carboplatin) will be administered for the first 4 cycles only, following Pemetrexed administration. If selected by the Investigator, Cisplatin (75 mg/m2) will be administered via IV infusion (approximately 30 minutes after pemetrexed infusion) Q3W for the first 4 cycles. If selected by the Investigator, Carboplatin will be administered at area under the concentration-time curve 5 mg/mL/min (AUC 5 mg/mL/min) Q3W immediately following the pemetrexed infusion for 4 cycles. Study Participants who meet eligibility criteria will be randomized in a 1:1 ratio intervention into the dostarlimab plus chemotherapy arm or the pembrolizumab plus Assignment chemotherapy arm, such that approximately 120 evaluable participants in each of the 2 arms complete the study. The randomization will be stratified by PD-L1 status of the tumor (TPS <1% vs 1% to 49% vs ≥50%) and smoking status (never vs former/current).



#### 2. STATISTICAL HYPOTHESES

The primary efficacy endpoint, ORR using RECIST v1.1 based on BICR, of dostarlimab plus chemotherapy is similar to that of pembrolizumab plus chemotherapy in participants with metastatic non-squamous NSCLC without a known EGFR, ALK, ROS-1, or BRAF V600E mutation or other genomic aberration for which an approved targeted therapy is available and who have not received prior treatment of metastatic disease.

#### 2.1. Multiplicity Adjustment



# 3. ANALYSIS SETS

The analysis sets are presented in Table 4.

Table 3 Analysis Sets





#### 4. STATISTICAL ANALYSES

#### 4.1. General Considerations

#### 4.1.1. General Methodology

The ITT Set will be used for all Study Population analyses and Efficacy analyses and the Safety Analysis Set will be used for all safety analyses, unless otherwise stated.

Analysis and summaries performed on the ITT set will be presented by treatment assigned to the participant during randomization unless otherwise specified.

#### 4.1.2. Baseline Definition



#### 4.1.3. Multicenter Studies

In this multicenter global study, enrolment will be presented by country and site.



#### 4.1.4. Visit Windows

It is expected that all visits should occur according to the protocol schedule.

#### 4.1.5. Study Population Summaries

The OPS document will provide additional details regarding the participant disposition and study population summaries, including, but not limited to the following:

- Participant status and disposition
- Treatment status and reasons for discontinuation of study treatment
- Screen status and reasons for screen failures
- Participants by country and site ID
- Important protocol deviations
- Study populations
- Demographics and baseline characteristics (including age, gender, ethnicity, race, and stratification factors: smoking status and PD-L1 status)
- Medical history / physical exam
- Advanced/Metastatic NSCLC history
- Prior anti-cancer therapy, prior radiotherapy and prior surgery
- Subsequent anti-cancer therapy
- Prior and concomitant medications
- Concomitant procedures

#### 4.2. Primary Endpoint Analyses

The primary efficacy endpoint objective response rate (ORR) will be evaluated by RECIST v1.1 based on blinded independent central review (BICR). The primary analysis of ORR will be based on the ITT population, and a supportive sensitivity analysis will be performed on the response evaluable population and per-protocol population.



#### 4.2.1. Definition of endpoint

ORR per RECIST v1.1 is defined as the proportion of patients who have a complete response (CR) or partial response (PR) as their best overall response (BOR) based on BICR.

Best Overall Response (BOR)

The best overall response is the best response recorded from the date of randomization until disease progression or initiation of new anti-cancer therapy, whichever is earlier, as assessed by the BICR per RECIST v1.1, using all scans regardless of whether they were scheduled or not. The order from best to worst of the available responses is CR, PR, stable disease (SD), progressive disease (PD) and not evaluable (NE). In order to assign a BOR of CR or PR, a participant initial response must be confirmed by repeat assessment performed no less than 4 weeks after the initial criteria for response were met.



#### 4.2.2. Main analytical approach





#### 4.2.3. Sensitivity analyses



# 4.3. Secondary Endpoints Analyses

The secondary efficacy endpoints overall survival (OS) and progression free survival (PFS) using RECIST v1.1 based on Investigator assessment will be evaluated. They will be summarized using the ITT population.

#### 4.3.1. Definition of endpoints

#### 4.3.1.1. Overall Survival (OS)

Overall Survival (OS), defined as the interval of time (in months) from randomization to the date of death due to any cause, regardless of whether the patient withdraws from randomized therapy or receives another anti-cancer therapy.



#### 4.3.1.2. Progression-Free Survival per RECIST v1.1 (PFS)

Progression-free survival (PFS) per RECIST v1.1 based on investigator assessment, defined as the interval of time (in months) between the date of randomization and the earlier of the date of disease progression (PD) as assessed by the investigator per RECIST 1.1 criteria and the date of death due to any cause.



Determination of dates of PFS events and dates for censoring are described in Table 4.





- 4.3.2. Main analytical approach
- 4.3.2.1. Overall Survival (OS)



4.3.2.2. Progression-Free Survival per RECIST v1.1 (PFS)

| CCI |
|-----|



## 4.4. Supportive Secondary Endpoint(s)

#### 4.4.1. Adverse Events/Serious Adverse Events

The safety analyses will be based on the Safety Analysis Set, unless otherwise specified.









# 4.5. Exploratory Endpoints Analyses



| CCI |
|-----|



















# 4.6. Other Analyses





# 4.7. Interim Analyses

No formal interim analysis is planned for this study.

# 4.8. Changes to Protocol Defined Analyses

Changes from the originally planned statistical analysis specified in the protocol amendment 5 (Dated: 14-FEB-2023) are outlined below.

| Pro | tocol | Statistical Analysis Plan | Rationale for Changes |
|---|---|---|---|
| • | No formal interim analysis will be done for this study. | CCI | CCI |
| • | There is no protocol defined adverse events of special interest (AESI) for Dostarlimab. | Analyses of AESIs are<br>based on pre-defined<br>MedDRA PTs. | CCI |

| Protocol | Statistical Analysis Plan | Rationale for Changes |
|----------|---------------------------|-----------------------|
| | | CCI |
| CCI | | |

# 5. SAMPLE SIZE DETERMINATION



# 6. SUPPORTING DOCUMENTATION

# 6.1. Appendix 1 Abbreviations and Trademarks

# 6.1.1. List of Abbreviations

| Abbreviation | Description |
|--------------|------------------------------------------------|
| CCI | |
| AE | Adverse Event |
| AESI | Adverse Event of Special Interest |
| ALT | Alanine Aminotransferase |
| BICR | Blinded Independent Central Review |
| BoR | Best Overall Response |
| CI | Confidence Interval |
| CCI | |
| CR | Complete Response |
| CTCAE | Common Terminology Criteria for Adverse Events |
| CCI | |
| DCO | Data Cut-Off |
| DCR | Disease Control Rate |
| CCI | |

| Abbreviation | Description |
|--------------|----------------------------------------------|
| ECG | Electrocardiogram |
| ECOG | Eastern Cooperative Oncology Group |
| eCRF | Electronic Case Record Form |
| EGFR | Epidermal Growth Factor Receptor |
| CCI | Epidermar Growth Factor Receptor |
| GSK | GlaxoSmithKline |
| HR | Hazard Ratio |
| CCI | |
| CCI | |
| irAE | Immune Related Adverse Event |
| ITT | Intent-To-Treat |
| MedDRA | Medical Dictionary for Regulatory Affairs |
| NE | Not Evaluable |
| NQ | Non-quantifiable |
| NSCLC | Non-Small Cell Lung Cancer |
| OPS | Output and Programming Specification |
| ORR | Objective Response Rate |
| OS | Overall Survival |
| PCI | Potential Clinical Importance |
| PD | Progressive Disease |
| CCI | |
| PFS | Progression Free Survival |
| CCI | |
| PP | Per-Protocol |
| PR | Partial Response |
| CCI | |
| PT | Preferred Term |
| QTc | QT Interval Corrected for Heart Rate |
| Q3W | Every Three Weeks |
| RECIST CCI | Response Evaluation Criteria in Solid Tumors |
| SAP | Statistical Analysis Plan |
| SAE | Serious Adverse Event |
| SD | Stable Disease |
| SMQ | Standardized MedDRA Query |
| SOC | System Order Class |

| Abbreviation | Description |
|--------------|----------------------------------|
| TEAE | Treatment Emergent Adverse Event |
| TOI | Term of Interest |
| CCI | |
| ULN | Upper Limit of Normal |

#### 6.1.2. Trademarks

| Trademarks of the GlaxoSmithKline Group | Trademarks not owned by the |
|---|---|
| of Companies | GlaxoSmithKline Group of Companies |
| None | MedDRA |

# 6.2. Appendix 2: Exclusions from Per Protocol Population

The per-protocol population include all participants in the ITT who do not have protocol deviations that may significantly impact the interpretation of efficacy results.





# 7. REFERENCES

